CLINICAL TRIAL: NCT06606275
Title: The Safety and Effectiveness of Warfarin Vs Apixaban in Patients with Non-Valvular Atrial Fibrillation/ Venous Thromboembolism and End-Stage Kidney Disease on Dialysis
Brief Title: The Safety and Effectiveness of Warfarin Vs Apixaban in Patients with NVAF/ VTE and ESKD on Dialysis
Acronym: WARD
Status: Completed | Type: Observational
Sponsor: Abu Dhabi Health Services Company (Other Government)
Collaborators: United Arab Emirates University (Other); Cleveland Clinic Abu Dhabi (Other)
Responsible Party: Principal Investigator, Said Nabil, Clinical Pharmacist, Abu Dhabi Health Services Company
Other Study IDs: KD/AJ/1063
Record Dates: First submitted 2024-09-12; First posted 2024-09-20 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: End-Stage Kidney Disease (ESKD); Non-valvular Atrial Fibrillation (NVAF); Venous Thromboembolism (VTE)
Keywords: Warfarin; Apaxiban
MeSH Terms: conditions — Kidney Failure, Chronic; Venous Thromboembolism | interventions — apixaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Apixaban arm: Patient who were receiving warfarin while on dialysis
  Interventions: Drug: Apixaban
- Warfarin arm: Patient who were receiving warfarin while on dialysis
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Apixaban — Apixaban is a direct oral anticoagulant (DOAC) that inhibits factor Xa, playing a crucial role in preventing blood clot formation. It is commonly prescribed for stroke prevention in patients with non-valvular atrial fibrillation (NVAF) and for treating and preventing venous thromboembolism (VTE), including deep vein thrombosis (DVT) and pulmonary embolism (PE).
  Groups: Apixaban arm
Drug: Warfarin — Warfarin is a vitamin K antagonist widely used as an anticoagulant to prevent thromboembolic events, particularly in conditions like atrial fibrillation, venous thromboembolism, and in patients with mechanical heart valves. It inhibits the enzyme vitamin K epoxide reductase, thereby reducing the activation of vitamin K-dependent clotting factors (II, VII, IX, X) and regulatory proteins C and S. Due to its narrow therapeutic index, warfarin requires regular monitoring of the International Normalized Ratio (INR) to optimize anticoagulation while minimizing the risk of bleeding. Warfarin's pharmacokinetics and pharmacodynamics can be influenced by genetic polymorphisms, diet, and drug interactions, necessitating individualized dosing strategies.
  Groups: Warfarin arm

SUMMARY:
This is a retrospective study of End-Stage Kidney Disease (ESKD) patients on dialysis receiving apixaban or warfarin at Tawam Hospital [a tertiary care hospital in Al Ain, UAE]. The study aims to assess the appropriateness of prescribing apixaban and warfarin in this population and evaluate their safety and effectiveness.

DETAILED DESCRIPTION:
Direct oral anticoagulants (DOACs), including apixaban, are used for stroke prevention in non-valvular atrial fibrillation (NVAF) and for venous thromboembolism (VTE) management. Patients with end-stage kidney disease (ESKD) on dialysis face elevated risks of thromboembolic events and bleeding. While apixaban is FDA-approved for use in this population, its safety and efficacy compared to warfarin are not well established in this vulnerable population.

This retrospective observational study aims to assess the prescribing appropriateness of apixaban compared to warfarin and evaluate their safety and effectiveness in a cohort of ESKD patients undergoing dialysis. This study will include ESKD patients on dialysis receiving apixaban or warfarin at Tawam Hospital from May 1, 2018, to January 31, 2024. Data on demographics, anticoagulant dosing, therapy duration, bleeding events, CHA2DS2-VASc score, HAS-BLED score, and thromboembolic events will be collected. Safety will be assessed by bleeding incidents, and effectiveness will be measured by VTE and stroke events. Dose appropriateness was evaluated according to FDA guidelines for apixaban and INR targets for warfarin. Data will be collected for eligible patients through electronic medical records (EMR).

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18
* CKD on dialysis for at least 1 month
* NVAF or VTE
* On Apixaban or Warfarin for at least 1 month

Exclusion Criteria:

* Age less than 18
* Received dialysis for less than 1 month (i.e., were treated with dialysis for acute kidney injury).
* On Apixaban or Warfarin for less than 1 month
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-pregnant Adult (≥ 18 years), CKD-on-dialysis patients receiving Apixaban or Warfarin for at least 1 month
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From date of enrollment until the date of first bleeding event or date of death from any cause, whichever came first, assessed up to 6 months
  Safety will be assessed by Major/Minor bleeding incidents based on International Society on Thrombosis and Haemostasis (ISTH) criteria
Effectiveness: VTE | From date of enrollment until the date of first documented VTE event or date of death from any cause, whichever came first, assessed up to 6 months
  Effectiveness will be measured by VTE events based on documented radiography and/or wells score for PE/DVT
Effectiveness: Stroke | From date of enrollment until the date of first documented Stroke event or date of death from any cause, whichever came first, assessed up to 6 months
  The primary outcome is the occurrence of stroke events in the study population, confirmed through clinical evaluation (e.g., neurological assessment) and imaging (CT or MRI). Data will be collected and reported as the number of patients experiencing stroke events during the study period. The incidence will be further categorized by stroke type (ischemic or hemorrhagic) and the severity of the event, using the National Institutes of Health Stroke Scale (NIHSS) for assessment. Aggregated data will include the total number of stroke events, time to occurrence, and any associated patient outcomes (e.g., mortality, disability).

SECONDARY OUTCOMES:
Dose appropriateness | Up to 6 months
  This measure will evaluate the dose appropriateness of apixaban and warfarin in patients with end-stage kidney disease (ESKD) on dialysis. For apixaban, dose appropriateness will be assessed based on FDA dosing guidelines for patients with renal impairment, including dosage adjustments for specific clinical factors (e.g., age, weight, and concurrent medications). For warfarin, dose appropriateness will be evaluated using the target International Normalized Ratio (INR) range for stroke prevention or VTE management. The data will be aggregated and reported as the number and percentage of patients receiving guideline-concordant doses. In cases where dosing is not appropriate, discrepancies will be documented and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Mosab Albalas, PharmD, Study Director — Tawam Hospital; Said Nabil, MS, PharmD, Principal Investigator — Abu Dhabi Health Services Co. SEHA
Locations (1):
- SEHA Tawam Hospital, Al Ain City, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelly DM, Ademi Z, Doehner W, Lip GYH, Mark P, Toyoda K, Wong CX, Sarnak M, Cheung M, Herzog CA, Johansen KL, Reinecke H, Sood MM. Chronic Kidney Disease and Cerebrovascular Disease: Consensus and Guidance From a KDIGO Controversies Conference. Stroke. 2021 Jul;52(7):e328-e346. doi: 10.1161/STROKEAHA.120.029680. Epub 2021 Jun 3. PMID 34078109
- [Background] Christiansen CF, Schmidt M, Lamberg AL, Horvath-Puho E, Baron JA, Jespersen B, Sorensen HT. Kidney disease and risk of venous thromboembolism: a nationwide population-based case-control study. J Thromb Haemost. 2014 Sep;12(9):1449-54. doi: 10.1111/jth.12652. Epub 2014 Jul 29. PMID 25040558
- [Background] Cheung CYS, Parikh J, Farrell A, Lefebvre M, Summa-Sorgini C, Battistella M. Direct Oral Anticoagulant Use in Chronic Kidney Disease and Dialysis Patients With Venous Thromboembolism: A Systematic Review of Thrombosis and Bleeding Outcomes. Ann Pharmacother. 2021 Jun;55(6):711-722. doi: 10.1177/1060028020967635. Epub 2020 Oct 19. PMID 33073581
- [Background] Chen A, Stecker E, A Warden B. Direct Oral Anticoagulant Use: A Practical Guide to Common Clinical Challenges. J Am Heart Assoc. 2020 Jul 7;9(13):e017559. doi: 10.1161/JAHA.120.017559. Epub 2020 Jun 15. PMID 32538234
- [Background] Chen HY, Ou SH, Huang CW, Lee PT, Chou KJ, Lin PC, Su YC. Efficacy and Safety of Direct Oral Anticoagulants vs Warfarin in Patients with Chronic Kidney Disease and Dialysis Patients: A Systematic Review and Meta-Analysis. Clin Drug Investig. 2021 Apr;41(4):341-351. doi: 10.1007/s40261-021-01016-7. Epub 2021 Mar 11. PMID 33709339